CLINICAL TRIAL: NCT01639768
Title: A Randomized, Double-blind, Placebo-controlled Study to Determine Safety, Tolerability and the Optimal Effective Dose of SUBLIVAC FIX Birch in Patients With Allergic Rhinitis/Rhinoconjunctivitis Caused by Birch Pollen
Brief Title: SUBLIVAC FIX Birch Dose Tolerability/Dose Range Finding
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: HAL Allergy (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SB/0038
Record Dates: First submitted 2012-07-03; First posted 2012-07-13 (Estimated); Last update posted 2013-05-29 (Estimated); Status verified 2013-05

CONDITIONS: Allergic Rhinitis; Allergic Rhinoconjunctivitis
Keywords: Sublingual immunotherapy; Dose range finding; Dose tolerability; Birch pollen; Allergic rhinitis/rhinoconjunctivitis; Safety; Immunogenicity
MeSH Terms: conditions — Rhinitis, Allergic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- SUBLIVAC FIX Birch 0 AUN/ml (Placebo Comparator)
  Interventions: Drug: SUBLIVAC FIX Birch
- SUBLIVAC FIX Birch 3,333 AUN/ml (Active Comparator)
  Interventions: Drug: SUBLIVAC FIX Birch
- SUBLIVAC FIX Birch 10,000 AUN/ml (Active Comparator)
  Interventions: Drug: SUBLIVAC FIX Birch
- SUBLIVAC FIX Birch 20,000 AUN/ml (Active Comparator): Evaluation of the SUBLIVAC FIX Birch 20,000 AUN/ml by an independent safety committee
  Interventions: Drug: SUBLIVAC FIX Birch
- SUBLIVAC FIX Birch 40,000 AUN/ml (Active Comparator): Start of SUBLIVAC FIX Birch 40,000 AUN/ml arm depends on safety in the SUBLIVAC FIX Birch 20,000 AUN/ml arm evaluated by an independent safety committee
  Interventions: Drug: SUBLIVAC FIX Birch

INTERVENTIONS:
Drug: SUBLIVAC FIX Birch — Comparison of different dosages to placebo

SUMMARY:
The aim of the study is to determine the optimal effective dose of SUBLIVAC FIX Birch based on reduction of upper airways reactivity after 5 months of treatment with different dosages of SUBLIVAC FIX Birch compared to placebo. Furthermore, safety and tolerability will be assessed by the number of related Adverse Events of different dosages of SUBLIVAC FIX Birch compared to placebo.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent
* Age ≥ 18 ≤ 60 years
* Allergic rhinitis/rhinoconjunctivitis related to birch pollen with or without concomitant mild to moderate persistent asthma
* FEV1 > 70% for patients with a history of asthma, FEV > 70% or PEF > 80% for patients without a history of asthma
* A positive SPT (mean wheal diameter ≥ 3mm compared to negative control and negative control should be negative) for birch pollen assessed within

  1 year before randomization.
* Positive serum specific anti-birch IgE-test (> 0.7 U/mL)
* A positive TNPT for birch pollen at screening (Lebel score ≥ 6) at

  * 10,000 AU/mL

Exclusion Criteria:

* Patients with (expected) clinically relevant symptoms during the course of the trial due to concomitant sensitization i.e. positive SPT (mean wheal diameter ≥ 3mm) to allergens other than birch pollen
* Patients sensitized to pets should not be included if they are regularly exposed to pets and are symptomatic upon exposure to pets
* Completed immunotherapy (SCIT or SLIT) with birch pollen allergens within the past 5 years
* Completed unsuccessful specific immunotherapy in the past
* Vaccination within one week before start of therapy or during the initiation phase
* Anti-IgE therapy within the 6 months prior to inclusion and during the study
* Severe immune disorders (including auto-immune diseases) and/or diseases requiring immunosuppressive drugs
* Active malignancies or any malignant disease during the previous 5 years
* Severe uncontrolled diseases that could increase the risk for patients participating in the study, including but not limited to: cardiovascular insufficiency, any severe or unstable lung diseases, endocrine diseases, clinically significant renal or hepatic diseases, or haematological disorders
* Active inflammation or infection of the target organs (nose, eyes or lower airways) at the start of the study
* Moderate to severe nasal obstructive diseases that preclude a TNPT (septal deviation, nasal polyps, recent nasal surgery, etc.)
* Diseases with a contraindication for the use of Adrenaline (e.g. hyperthyroidism, glaucoma)
* Use of systemic steroids within 4 weeks before start of the study and during the study
* Treatment with systemic and local β-blockers
* Participation in a clinical study with a new investigational drug within the last 3 months or for a biological within the last 6 months prior to or during the study
* Pregnancy, lactation or inadequate contraceptive measures for women of child-bearing age (adequate contraceptive measures will be the use of a contraceptive device or -pill)
* Alcohol, drug or medication abuse within the past year
* Any clinically significant abnormal laboratory parameter at screening
* Lack of cooperation or compliance
* Severe psychiatric, psychological, or neurological disorders
* Patients who are employees of the institution or 1st grade relatives or partners of the investigator

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 270 (Actual)
Dates: Start 2012-07; Primary Completion 2013-03 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
Nasal Provocation Test (NPT) | 5 months
Number of related AEs | First ten days of study medication intake

SECONDARY OUTCOMES:
Serum specific immunoglobulin levels (IgE, IgG, IgG4) | 5 months
Number of local and systemic reactions | Duration of study medication intake (approximately 5 months)
Peak Nasal Inspiratory Flow (PNIF) | 5 months

CONTACTS AND LOCATIONS:
Overall Officials: Oliver Pfaar, PD. Dr. med., Study Chair — Zentrum für Rhinologie und Allergologie, An-den-Quellen-10, 65189 Wiesbaden, Germany
Locations (20):
- Czechia (5):
  - AKI, spol s. r.o., Brno
  - Ordinace Alergologie, Most
  - Respiral s. r.o., Pilsen
  - Ústav imunologie a alergologie, Pilsen
  - Kasmed s. r.o., Tábor
- Germany (3):
  - Praxis für Atemwegserkrankungen, Leipzig, Saxony
  - Medizinische Fakultät. Klinik und Poliklinik für HNO-Klinik, Dresden
  - HNO-Wiesbaden - Center for Rhinology and Allergology, Wiesbaden
- Poland (12):
  - Prywatna Praktyka Lekarska Gabinet Pediatryczno-Alergologiczny, Bialystok
  - NZOS "Zdrowie", Cieszyn
  - Poradnia Alergologiczna Samodzielnego Publicznego Szpitala Nr 5 Slaskiego Uniwersytetu Medycznego w Katowicach, Katowice
  - Specjalistyczny Ośrodek Alergologiczno-Internistyczny "ALL-MED", Krakow
  - Poradnia Alergologii i Chorób Płuc SP ZOZ Uniwersytecki Szpital Kliniczny Nr.1 im. Norberta Barlickiego w Łodzi, Lodz
  - NZOZ Centrum Alergologii, Lodz
  - ALERGOPNEUMA Marek Michnar i Wspolnicy Sp. Jawna, Lublin
  - NZOZ Centrum Alergologii, Lublin
  - Centrum Alergologii Teresa Hofman, Poznan
  - ALERGOMED Specjalistyczna Przychodnia Lekarska Sp. z o.o., Tarnów
  - EMC Intytut Medyczny S.A. Przychodnia przy Łowieckiej, Wroclaw
  - NZOZ Lekarze Specjaliści J. Małolepszy i Partnerzy, Wroclaw

REFERENCES:
- [Derived] Pfaar O, van Twuijver E, Boot JD, Opstelten DJ, Klimek L, van Ree R, Diamant Z, Kuna P, Panzner P. A randomized DBPC trial to determine the optimal effective and safe dose of a SLIT-birch pollen extract for the treatment of allergic rhinitis: results of a phase II study. Allergy. 2016 Jan;71(1):99-107. doi: 10.1111/all.12760. Epub 2015 Oct 26. PMID 26417901